CLINICAL TRIAL: NCT00748462
Title: Clinical Quality Assurance Study: Fractional CO2 Treatment of Acne Scars in Asians
Brief Title: Fractional CO2 Treatment of Acne Scars in Asians
Acronym: CO2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Woraphong Manuskiatti, M.D., Professor, Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SiEC 145/2551 (EC4); 1CIP7978- A02
Record Dates: First submitted 2008-07-01; First posted 2008-09-08 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Acne Scar, Wrinkle
Keywords: Acne scar, Wrinkle, Pigmentation, Fractional CO2 laser

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Fractional CO2 laser resurfacing
  Interventions: Device: Fractional CO2 Laser

INTERVENTIONS:
Device: Fractional CO2 Laser — the treatment settings:
  1. Pulse duration : 5 to 7ms depending on skin reaction
  2. Spot Density: 49 MTZ/cm2 (Low density)
  3. Power: 15 W = (75 - 105) mJ/MTZ
  Other Names: Juvia (trade mark)Fractional CO2 Laser

SUMMARY:
The objective of this study is to investigate the efficacy and side effects of a fractional CO2 laser for treatment of acne scar in Asians.

DETAILED DESCRIPTION:
* The objective of this study is to investigate the efficacy and side effects of a fractional CO2 laser for treatment of acne scar in Asians.
* Study hypothesis

  1. Reduction in acne scars based on blinded evaluation of before photos and the one and three month follow-up photos after four full face Ellipse Juvia with low density treatments with a fluency of 90-105 mJ/MTZ is statistically significant (5%).
  2. The direct clinical blinded evaluated reduction in acne scars based on before photos and the patient in life, by the one and three month follow-up is statistically significant (5%)
  3. Reduction in fine lines based on blinded evaluation of before photos and the one and three month follow-up photos after four full face Ellipse Juvia with low density treatments with a fluency of 90-105 mJ/MTZ is statistically significant (5%).
  4. The direct clinical blinded evaluated reduction in fine lines based on before photos and the patient in life, by the one and three month follow-up is statistically significant (5%).
  5. Reduction in pigmented disorders based on blinded evaluation of before photos and the one and three month follow-up photos after four full face Ellipse Juvia with low density treatments with a fluency of 90-105 mJ/MTZ is statistically significant (5%).
  6. The direct clinical blinded evaluated reduction in pigmented disorders based on before photos and the patient in life, by the one and three month follow-up is statistically significant (5%).
  7. Improvements in skin texture and pore size based on blinded evaluation of before photos and the one and three month follow-up photos after four full face Ellipse Juvia with low density treatments with a fluency of 90-105 mJ/MTZ is statistically significant (5%).
  8. The direct clinical blinded evaluated reduction in skin texture and pore size based on before photos and the patient in life, by the one and three month follow-up is statistically significant (5%).

ELIGIBILITY:
Inclusion Criteria:

* Numbers of volunteers: 10 healthy men and women
* Aged at least 30 year old
* Skin type: 1 - 4
* Degree of suntan: None - light
* Skin condition: visible acne scars

Exclusion Criteria:

* Fitzpatrick skin types 5-6.
* Patients with lesions with any clinical suspicion of being pre-cancerous or skin malignancies of any kind.
* Patients with skin diseases associated with Koebner phenomena.
* Patients who have used Botox or filler injection to the periorbital or perioral regions 12 months prior or during the study.
* Patients who have used topical retinoids, AHA under prescription or Vitamin C, 3 months prior to or during the study.
* Patients who are pregnant or who wish to become pregnant and lactating women.
* Patients who have been exposed to sun within 2 week from date of treatment.
* Patients prone to hypertrophic scars or keloids
* Patients who have previously undergone laser resurfacing may not be suitable for yet another procedure.
* Patients undergoing oral retinoid therapy for acne in the past 6 months.
* Patients who suffer from any serious medical condition, including diabetes, bleeding diathesis, delayed wound healing or prednisolone intake.
* Patients with wound infections (herpes, other) on the day of treatment.
* Patients with moderate and severe inflammatory acne, Immunosuppressed patients, History of vitiligo.
* Patients with unrealistic concerns/expectations and inability to do the appropriate post-operative care.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
by the clinical investigator and graded into one of six categories: worse, no effect, slightly better, fair, good, and excellent. The results shall be reported. | Follow-up 1 and 3 months after the last treatment

SECONDARY OUTCOMES:
The outcome and degree of satisfaction based on the before photo is evaluated by the patients themselves | Follow-up 1 and 3 months after the last treatment

CONTACTS AND LOCATIONS:
Overall Officials: Woraphong Manuskiatti, M.D., Principal Investigator — Department of Dermatology, Siriraj Hospital
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand

REFERENCES:
- [Background] Fitzpatrick RE. Laser resurfacing today and the "cookbook" approach: a recipe for disaster? A comment. J Cosmet Dermatol. 2005 Dec;4(4):298-9; author reply 299-300. doi: 10.1111/j.1473-2165.2005.00208.x. No abstract available. PMID 17168879
- [Background] Fitzpatrick RE, Goldman MP, Satur NM, Tope WD. Pulsed carbon dioxide laser resurfacing of photo-aged facial skin. Arch Dermatol. 1996 Apr;132(4):395-402. PMID 8629842
- [Background] Alster TS, Lupton JR. Erbium:YAG cutaneous laser resurfacing. Dermatol Clin. 2001 Jul;19(3):453-66. doi: 10.1016/s0733-8635(05)70286-2. PMID 11599402
- [Background] Manstein D, Herron GS, Sink RK, Tanner H, Anderson RR. Fractional photothermolysis: a new concept for cutaneous remodeling using microscopic patterns of thermal injury. Lasers Surg Med. 2004;34(5):426-38. doi: 10.1002/lsm.20048. PMID 15216537